CLINICAL TRIAL: NCT04683562
Title: The Implication of Placental Netrin-1 Receptor DCC in the Pathophysiology of Placenta Accreta
Brief Title: Netrin-1 and Placenta Accreta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PA-NT1
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal pregnancy group (Other)
  Interventions: Other: Pregnant women at 28-32 weeks; Other: at delivery
- Placenta accreta group (Other)
  Interventions: Other: Pregnant women at 28-32 weeks; Other: at delivery

INTERVENTIONS:
Other: Pregnant women at 28-32 weeks — Pregnant women at gestational age 28-32 weeks
Other: at delivery — women delivered at term

SUMMARY:
Netrin-1 is a secreted protein, which was first identified as a neuronal guidance factor. It is expressed in a multitude of tissues as pancreas, lung, breast, and placenta. Netrin-1 is a multifunctional protein, involved in cell polarity, adhesion, angiogenesis, apoptosis, migration, morphogenesis, and differentiation of various cell types. Most of netrin-1 activity occur through signaling pathways induced by its two main receptors, DCC (deleted in colorectal cancer) and UNC5H (uncoordinated-5 homolog). Its receptors have been linked to the processes of apoptosis and angiogenesis. In absence of netrin-1, DCC and UNC5H receptors lead to apoptosis. In contrary, in presence of netrin-1, receptors transduce molecular cascades leading to proliferation, differentiation and migration of the cells. Netrin-1 has been involved in the pathogenesis of multiple diseases, as diabetes, cardiovascular diseases, and cancer. Serum Netrin-1 levels were high in preeclamptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-40 years.
* Singleton pregnancy.
* Women with suspicion of PA by two-dimensional (2D) gray scale imaging and color Doppler flow mapping

Exclusion Criteria:

* Multiple pregnancy,
* Fetal anomalies,
* Preterm premature rupture of membranes, or infection
* Any medical disorders, such as thyroid dysfunction, hypertension, and gestational diabetes
* Patients with known bleeding disorders or on anticoagulant therapy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Placental Netrin-1 level | 4 weeks
  will be measured by using enzyme-linked immunosorbent assay (ELİSA) in placental homogenate

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided